CLINICAL TRIAL: NCT06648447
Title: Investigation of the Efficacy and Tolerability of Topical Applied Tirbanibulin on Actinic Keratoses With Downward-directed Proliferation Patterns
Acronym: Tir2401
Status: Recruiting | Type: Observational
Sponsor: Thomas Dirschka (Network)
Responsible Party: Sponsor-Investigator, Thomas Dirschka, Clinical Professor, CentroDerm GmbH
Organization: CentroDerm GmbH (Network)
Other Study IDs: CentroDerm_TIR24001
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Actinic Keratosis (AK)
Keywords: actinic keratosis; klisyri; tirbanibulin; proliferating actinic keratosis; proliferating actinic keratoses; LC-OCT
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 70 Days
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The aim of this study is to observe the influence of tirbanibulin on proliferation patterns of actinic keratoses (efficacy on proliferation score according to Schmitz et al.). For this purpose, tirbanibulin is applied in-label, proliferation is measured by LC-OCT at different time points and dermatohistopathology is performed (optionally) at the end. Local skin reactions to the product will also be recorded (tolerability).

DETAILED DESCRIPTION:
Actinic keratoses (AK) are premalignant skin changes of a cutaneous squamous cell carcinoma (SCC), which are often triggered by UV exposure. Clinically, they appear as small, rough, reddish, sandpaper-like patches, occasionally also as hyperkeratotic lesions. They are one of the most common reasons for dermatological consultations, and their incidence has been steadily increasing in recent years due to changes in leisure habits with increased UV exposure and demographic changes in the population, such as those observed in Germany.

While the mortality rate of squamous cell carcinoma of the skin is low, the persistence and recurrence of AK, which requires frequent treatment, is a challenge for both patients and healthcare systems.

There are numerous treatment options for AK, ranging from surgical and cryosurgical interventions to ablative laser treatments, topical and photodynamic therapies. These treatments can generally be categorized as lesion- or field-oriented.

Some AK show resistance to conventional therapies. This could possibly be due to different proliferation patterns of AK. Schmitz et al. established the PRO score, an instrument that describes the proliferation behavior of AK in a three-stage scale. This histological score is well validated and is increasingly used in histological diagnostics. New imaging techniques such as confocal line-field optical coherence tomography (LC-OCT) enable real-time assessment of histological parameters without the need for biopsies. In LC-OCT it is possible to detect the PRO Score of an AK in a few seconds.

Clinical parameters such as the Olsen grade, on the other hand, record the visible or palpable hyperkeratosis of an AK. However, the significance of hyperkeratosis for the risk of progression of AK to SCC is only of minor importance. Histological diagnostics and LC-OCT therefore make it possible to determine this risk more precisely.

Similarly, clinical scores such as the Olsen garde do not indicate which AKs are refractory to therapy, and which respond to therapy. One reason for this could be the proliferation behavior of the individual AK. Tirbanibulin, which primarily targets this cell proliferation, is a promising agent for the treatment of highly proliferative AK (PRO II and III). One aim is to observe its effects on basal proliferation after treatment, which can be assessed in real time using LC-OCT. This non-invasive method provides rapid evaluations within minutes. In addition to efficacy in proliferative AK, evaluation of the tolerability of tirbanibulin is crucial to contextualize its role in therapy. It is therefore of interest to determine whether increased skin reactions in proliferative AK correlate with improved clearance rates.

Tirbanibulin is a method frequently used in practice for the treatment of actinic keratoses. The application is quick with only 5 consecutive applications, results in only a minor local reaction and is nevertheless effective. In this study, various parameters such as local tolerance, the Olsen grade and the PRO score will be monitored using LC-OCT. Patients with clinically confirmed AK for whom in-label therapy with tirbanibulin is planned anyway will be included.

ELIGIBILITY:
Inclusion Criteria:

* male, female, diverse patients (> 18yo) who are capable of giving consent
* female patients are eligible if the patient is not a woman of childbearing potential (WOCBP) or if she is postmenopausal (cessation of menstruation >12 months) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, total hysterectomy)
* signed informed consent
* diagnosis of at least 1 non-hypertrophic, non-hyperkeratotic actinic keratosis of the scalp or face with Olsen Grade I and PRO II or III
* planned treatment of AK with Klisyri® before study start and indepently of the study
* the study participant is in good general condition for his or her age and does not currently have any active diseases that, in the opinion of the investigator, justify exclusion from the study

Exclusion Criteria:

* known or documented intolerance to any of the ingredients of Klisyri®
* any planned AK treatment other than Klisyri® in the treatment area
* treatment of actinic keratoses in the treatment area within the past 3 Months (e.g. photodynamic therapy, topical 5-FU, diclofenac, imiquimod, cryotherapy etc.)
* suspected invasive squamous cell cancer in the treatment area
* chronic wounds, erosions, pre-existing inflamed or infected skin with disruption of the epidermal barrier in the treatment area
* suspected non-compliance
* current or within the last 8 weeks given systemic cancer medication
* any other topical treatment against actinic keratosis in the treatment area within the past 12 weeks
* any contraindication according to the Summary of Product Characteristics (SmPC) of Klisyri®
* any systemic immunosuppressant given within the 8 weeks prior to the study (e.g. systemic prednisolone, azathioprine etc.)
* locally applied retinoids, steroids, or other prescribed externals in the 4 weeks prior to the start of the study in the treatment area that, in the opinion of the study physician, necessitate exclusion
* products containing glycolic or alpha-hydroxy acids applied locally in the treatment area in the last 4 weeks
* chemical peelings in the treatment area in the last 4 weeks
* simultaneous participation in a clinical trial
* participation in a clinical study within the last 30 days
* family members or colleagues of the investigator or the investigational team or the CRO
* patient is in a position or has a relationship with the investigator that presents a potential conflict of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the medical office (Berufsausübungsgemeinschaft Prof. Dr. Dirschka und Priv.-Doz. Dr. Schmitz).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
- Improvement of the PRO score of the marker lesion at D57 (LC-OCT) and/or clearance in LC-OCT of marker lesion at D57 | 70 days after inclusion (57 days after visit 2)
  Measurement will be done by LC-OCT to detect the PRO Score of the actinic keratosis.
assessment of local skin reaction grading scale at V2 | 14 days after baseline visit
  Assessment of the local skin reaction via a 4-point-likert scaled measurement of erythema, scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration

SECONDARY OUTCOMES:
Clinical clearance of marker lesion at visit 2 | 14 days after baseline visit
  Clinical clearance of the previously marked actinic keratosis
Clinical clearance of marker lesion at visit 3 | 70 days after baseline
  Clinical clearance of predefined actinic keratosis at visit 3
Improvement of PRO Score at V2 | 14 days after baseline
  Improvement of PRO score at visit 2 in LC-OCT (line-field optical coherence tomography)
LC-OCT clearance of marker lesion at V2 | 14 days after baseline
  Clearance of marker lesion at visit 2 in LC-OCT (line-field optical coherence tomography)
Histopathological clearance of marker lesion at V3 | 70 days after baseline
  histopathological clearance of predefined AK at V3. Only applicable if histopathology was performed afterwards (in case of persisting AKs)

CONTACTS AND LOCATIONS:
Locations (1):
- CentroDerm, Wuppertal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No